CLINICAL TRIAL: NCT04687631
Title: Conversion Therapy of RAS/BRAF Wild-Type Colorectal Cancer Patients With Initially Unresectable Liver Metastases: mFOLFOXIRI Plus Cetuximab Versus mFOLFOXIRI Plus Bevacizumab
Brief Title: Conversion Therapy of RAS/BRAF Wild-Type Colorectal Cancer Patients With Initially Unresectable Liver Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Deputy director of the department of general surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRUST
Record Dates: First submitted 2020-12-27; First posted 2020-12-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: Cetuximab; Bevacizumab; Triplet Chemotherapeutic Regimen; Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOXIRI plus Cetuximab (Experimental)
  Interventions: Drug: mFOLFOXIRI plus Cetuximab
- mFOLFOXIRI plus Bevacizumab (Experimental)
  Interventions: Drug: mFOLFOXIRI Plus Bevacizumab

INTERVENTIONS:
Drug: mFOLFOXIRI plus Cetuximab — cetuximab 500mg/m2 + oxaliplatin 85 mg/m2 + irinotecan 165 mg/m2 + folinic acid 400 mg/m2 + 5-fluorouracil 2400 mg/m2 46h infusion starting on day 1, every 2 weeks
  Arms: mFOLFOXIRI plus Cetuximab
Drug: mFOLFOXIRI Plus Bevacizumab — bevacizumab 5mg/kg + oxaliplatin 85 mg/m2 + irinotecan 165 mg/m2 + folinic acid 400 mg/m2 + 5-fluorouracil 2400 mg/m2 46h infusion starting on day 1, every 2 weeks
  Arms: mFOLFOXIRI plus Bevacizumab

SUMMARY:
Evidence suggests that the addition of cetuximab or bevacizumab to doublet regimens could improve response rate and resectability rate of liver metastases and survival in colorectal liver metastases (CRLM). Moreover, it is observed that FOLFOXIRI yields higher response and resection rates compared with doublet regimens. However, which is better in conversion therapy of RAS/BRAF wild-type initially unresectable CRLM, FOLFOXIRI plus cetuximab or bevacizumab, remains unknown.

In this study, RAS/BRAF wild-type colorectal cancer patients with initially unresectable liver-only metastases, as prospectively confirmed by a local multidisciplinary team (MDT) according to predefined criteria, will be randomised between modified FOLFOXIRI (mFOLFOXIRI) plus cetuximab and mFOLFOXIRI plus bevacizumab. Patient imaging will be reviewed for resectability by MDT, consisting of at least one radiologist and three liver surgeons every assessment. MDT review will be performed prior to randomization as well as during treatment, as described in the protocol.

DETAILED DESCRIPTION:
Patients will be stratified for primary tumor location (right-sided or left sided) and numbers of liver metastases (<5 or ≥5).

Patients with RAS/BRAF wild-type primary tumors will be randomized between mFOLFOXIRI plus cetuximab (cetuximab 500 mg/m^2 in 60 minutes i.v., followed by oxaliplatin 85 mg/m^2 i.v. in 120 minutes, followed by irinotecan 165 mg/m^2 i.v. in 60 minutes, together with leucovorin 400 mg/m^2 i.v. in 120 minutes, followed by continuous infusion of 5-fluorouracil 2400 mg/m^2 in 46 hours, every 2 weeks) or mFOLFOXIRI plus bevacizumab (Bevacizumab 5 mg/kg in 15-30 minutes i.v., followed by oxaliplatin 85 mg/m^2 i.v. in 120 minutes, followed by irinotecan 165 mg/m^2 i.v. in 60 minutes, together with leucovorin 400 mg/m^2 i.v. in 120 minutes, followed by continuous infusion of 5-fluorouracil 2400 mg/m^2 in 46 hours, every 2 weeks).

Patients will be evaluated every 8 weeks by MRI or CT scan for disease status. The assigned systemic treatment should be continued for at least 6 months or earlier in case of resectability, progression of disease, unacceptable toxicity, or patient refusal. If after 6 months MDT concludes that the patient is still not resectable, it is highly unlikely that resectability will be achieved at all. Therefore the chemotherapy regimen may be reconsidered after 6 months of treatment.

In patients who will become resectable and undergo secondary surgery of liver metastases, the total duration of preoperative and postoperative treatment together should be 6 months. However, the postoperative chemotherapy regimen was determined by the investigator.

After 70% of patients were enrolled and conversion therapy were finished, a mid-term analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. The primary tumor was confirmed by histology as colorectal adenocarcinoma
2. Initially unresectable liver metastases suggested by MDT
3. RAS/BRAF gene wild-type states
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Life expectancy ≥ 3 months
6. Good hematological function: neutrophil ≥ 1.5x109 / L and platelet count ≥ 100x109 / L; HB ≥ 9g / dl (within one week before randomization)
7. Normal liver and kidney function: serum bilirubin ≤ 1.5x normal upper limit (ULN), alkaline phosphatase ≤ 5x ULN, serum transaminase (AST or ALT) ≤ 5x ULN (within one week before randomization);
8. Sign the written informed consent to participate in the experiment

Exclusion Criteria:

1. Patients with liver metastases from colorectal cancer who have previously received targeted therapy, chemotherapy, radiotherapy or interventional therapy
2. Known or suspected extrahepatic metastasis
3. Patients with known hypersensitivity to any component of the study treatment
4. Clinical related coronary heart disease or history of myocardial infarction in the last 12 months or left ventricular ejection fraction below normal range
5. Acute or subacute intestinal obstruction
6. Pregnancy (no pregnancy confirmed by serum / urine β - hCG) or breastfeeding.
7. Other malignant tumors within 5 years, except for those with skin basal cell carcinoma or cervical cancer
8. Known drug / alcohol abuse
9. No legal capacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Conversion resection rate of liver metastases | up to 6 months
  Rate of conversion from initially unresectable liver metastases to resectable ones

SECONDARY OUTCOMES:
Objective Response Rate | up to 6 months
  rate of objective response for therapy
Incidence of adverse events | up to 6 months
  Incidence of adverse events
Progression-Free Survival | up to 3 years
  Progression free survival
Overall Survival | up to 3 years
  overall survival
Early tumor shrinkage | at 8 weeks
  The rates of tumor shrinkage by RECIST at 8 weeks
Best deepness of response | up to 6 months
  the maximum tumor shrinkage rates by RECIST during the treatment of the study
time interval from chemotherapy to hepatectomy | up to 6 months
  Time interval from the beginning of treatment to hepatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, MD, Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No